CLINICAL TRIAL: NCT03547583
Title: A Randomized Parallel-group, Placebo-controlled, Double-blind, Multi-center Trial to Evaluate the Efficacy and Safety of the Oral sGC stImulator Vericiguat to Improve Physical Functioning in Activities of Daily Living in Patients With Heart Failure and Preserved Ejection Fraction (VITALITY-HFpEF)
Brief Title: Patient-reported Outcomes in Vericiguat-treated Patients With HFpEF
Acronym: VITALITY-HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Canadian VIGOUR Centre (Other); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19334; 2018-000298-65 (EudraCT Number)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-11

CONDITIONS: Chronic Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vericiguat up to 10 mg (Experimental): Subjects will receive vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, with sham titration at week 6.
  Interventions: Drug: Vericiguat (BAY1021189) 2.5 mg, 5 mg or 10 mg IR tablets
- Vericiguat up to 15 mg (Experimental): Subjects will receive vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, and to 15 mg at week 6.
  Interventions: Drug: Vericiguat (BAY1021189) 2.5 mg, 5 mg or 10 mg IR tablets
- Placebo (Placebo Comparator): Subject will receive placebo for 24 weeks, once daily, starting sham up-titration at weeks 2, 4, and 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) 2.5 mg, 5 mg or 10 mg IR tablets — Oral use. Vericiguat, which will be started at 2.5 mg at randomization and up-titrated to 5 mg at week 2, and to 10 mg at week 4, with sham titration or up-titration to 15 mg at week 6.
  Arms: Vericiguat up to 10 mg; Vericiguat up to 15 mg
Drug: Placebo — Placebo and sham up-titration at weeks 2, 4, and 6
  Arms: Placebo

SUMMARY:
The primary hypothesis in this trial is that the treatment with vericiguat 10 mg or 15 mg in patients with HFpEF improves the KCCQ PLS (Kansas City Cardiomyopathy Questionnaire Physical limitation score) compared to placebo after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of chronic heart failure (HF)
* HF decompensation within 6 months prior to randomization, defined as hospitalization for HF or intravenous (IV) diuretic treatment for HF without hospitalization.
* N-terminal pro brain natriuretic peptide (NT-proBNP) ≥300 or brain natriuretic peptide (BNP) ≥100 pg/mL in sinus rhythm, or NT-proBNP

  ≥600 or BNP ≥200 pg/mL in atrial fibrillation within 30 days prior to randomization
* Diagnostic criteria of HFpEF by echocardiography assessed within 12 months prior to randomization (most recent measurement must be used to determine eligibility with no interim event signaling potential deterioration in ejection fraction)

  * Left ventricular ejection fraction (LVEF) ≥45% and
  * Structural changes indicated by at least one of the following parameters:

    * Left ventricle (LV) hypertrophy (any of the following: intraventricular septal or posterior wall thickness ≥1.1 cm, and/or LV mass index ≥115 g/m*2 in male and ≥95 g/m*2 in female), or
    * Left atrium (LA) enlargement (any of the following: left atrial volume (LAV) index ≥29 ml/m*2, or LAV >58 mL in male and >52 mL in female patients, or LA area >20 cm*2, or LA diameter >40 mm in male and >38 mm in female patients)
* NYHA class II or III at randomization

Exclusion Criteria:

* Clinical instability at randomization, defined by

  * Any IV treatment within 24h prior to randomization, and/or
  * SBP ≥160 mmHg
  * SBP <110 mmHg and/or DBP <40 mmHg and/or symptomatic hypotension
  * Resting heart rate (HR) <50 or ≥100 beats per minute (bpm)
* Use of IV inotropes at any time between qualifying HF event and randomization
* Previous diagnosis of reduced ejection fraction (EF) (EF <40%)
* Hypertrophic obstructive cardiomyopathy, acute myocarditis, amyloidosis, sarcoidosis, or pericardial disease
* Primary valvular heart disease requiring surgery or intervention, or within 3 months after valvular surgery or intervention, or active endocarditis
* Acute coronary syndrome, including unstable angina, Non ST-elevation myocardial infarction or ST-elevation myocardial infarction, or Coronary artery bypass grafting (CABG) within 60 days prior to randomization, or indication for Percutaneous coronary intervention or CABG at the time of randomization
* Symptomatic carotid stenosis, or transient ischemic attack or stroke within 60 days prior to randomization
* Complex congenital heart disease
* Non-cardiac comorbidity (any of the following)

  * Estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m*2 calculated by Modification of Diet in Renal Disease formula
  * Hepatic insufficiency classified as Child-Pugh B or C
  * Morbid obesity with a body mass index >45 kg/m*2
  * Malignancy or other non-cardiac condition limiting life expectancy to <1 year, per physician judgment
  * Requires continuous home oxygen for severe pulmonary disease or has interstitial lung disease
  * Patients with allergies, intolerance or hypersensitivity to investigational drug or any of the excipients
* Concurrent or anticipated use of nitrates or NO donors, phosphodiesterase type V (PDE5) inhibitors, or a Soluble guanylate cyclase (sGC) stimulator

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (176):
- United States (29):
  - WestSide Medical, Beverly Hills, California
  - Capitol Interventional Cardiology, Carmichael, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Penrose-St. Francis Health Services, Colorado Springs, Colorado
  - Cardiology Associates of Fairfield County, PC, Trumbull, Connecticut
  - Cardiology Associates Of South Florida PA, Boynton Beach, Florida
  - Cardiovascular and Vein Center of Florida, Bradenton, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - LifeSpring Research Foundation, LLC, Miami, Florida
  - Southwest Florida Research, Naples, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - Cardiology Partners, Wellington, Florida
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Reid Health, Richmond, Indiana
  - Research Integrity, LLC, Owensboro, Kentucky
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Anne Arundel Health System, Annapolis, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Riser Medical Associates, Picayune, Mississippi
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Bryan Heart, Lincoln, Nebraska
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Corporation Lane Research Center, Virginia Beach, Virginia
- Argentina (8):
  - Clínica DIM, Ramos Mejía, Buenos Aires
  - Instituto de Investigaciones Clínicas San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Centro de Investigaciones Clínicas, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Centro de Medicina Integral e Investigacion Clínica, CABA, Ciudad Auton. de Buenos Aires
  - Centro de Especialidades Médicas, Villa Luro, Ciudad Auton. de Buenos Aires
  - Sanatorio Parque S.A., Rosario, Santa Fe Province
  - Inst. de Cardiología de Corrientes Juana Francisca Cabral, Corrientes
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Austria (7):
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Medizinische Universität Graz, Graz, Styria
  - Krankenhaus St. Josef Braunau, Braunau am Inn, Upper Austria
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Zentrum f. klinische Studien Dr. Hanusch GmbH, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Floridsdorf - Krankenhaus Nord, Vienna
- Belgium (5):
  - Algemeen Stedelijk Ziekenhuis Campus Aalst, Aalst
  - AZ St-Jan Brugge Oostende AV, Bruges
  - UZ Antwerpen, Edegem
  - H. Hartziekenhuis Mol, Mol
  - AZ Delta, Roeselare
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment Pazardzhik, Pazardzhik
  - Spec Hosp for Active Treatm in Cardiology Sv Georgi Pernik, Pernik
  - Specialized Hospital for Actrive Treatm of Card - Pleven, Pleven
  - Multiprofile Hospital for Active Treatment Medline Clinic, Plovdiv
  - MHAT Dr. Bratan Shukerov AD, Smolyan
  - Second Medical Center Sofia EOOD, Sofia
  - NMTH Tzar Boris III, Sofia
  - V MHAT, Sofia
  - MHAT Sveta Marina EAD, Varna
- Canada (10):
  - University of Alberta, Edmonton, Alberta
  - SMH Cardiology Clinical Trials Inc, Surrey, British Columbia
  - Cardiovascular CRO Ltd., Greater Sudbury, Ontario
  - London Health Sciences Centre, London, Ontario
  - PACE Cardiology Clinic, Newmarket, Ontario
  - Oakville Cardiologists, Inc., Oakville, Ontario
  - St. Michael's Hospital Health Centre, Toronto, Ontario
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Centre De Recherche Du (CRCHUM) - Hotel-Diu, Montreal, Quebec
  - CardioVasc HR, Inc., Saint-Jean-sur-Richelieu, Quebec
- Colombia (5):
  - Hospital General de Medellin, Medellín, Antioquia
  - IPS Centro Cientifico Asistencial S.A.S, Barranquilla, Atlántico
  - Caja de Compensación Familiar CAFAM, Bogotá, Bogota D.C.
  - Mediservis del Tolima IPS S.A.S, Ibagué, Tolima Department
  - Fundación Cardiovascular de Colombia, Floridablanca
- Germany (7):
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Zentrum für Klinische Studien Südbrandenburg GmbH, Elsterwerda, Brandenburg
  - Herz- und Diabeteszentrum Nordrhein-Westfalen (HDZ NRW), Bad Oeynhausen, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - St. Vincenz und Elisabeth Hospital, Kathol. Klinikum Mainz, Mainz, Rhineland-Palatinate
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Cardiologicum Hamburg - Praxen Wandsbek, Hamburg
- Greece (6):
  - KAT General Hospital of Athens, Kifisia / Athens, Attica
  - G. GENNIMATAS General State Hospital of Athens, Athens
  - University General Hospital of Larissa, Larissa
  - Konstantopoulio General Hospital of Nea Ionia - AGIA OLGA, Nea Ionia / Athens
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
- Hungary (5):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont Honvedkorhaz, Budapest
  - Pharma4Trial Kft., Gyöngyös
  - Kanizsai Dorottya Hospital, Nagykanizsa
  - Medifarma-98 Egeszsegugyi, Kereskedelmi es Szolgaltato Kft., Nyíregyháza
- Israel (9):
  - HaEmek Medical Center, Afula
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Corporation, Haifa
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Health Corporation of the Ziv Medical Center (R.A.), Safed
  - The Baruch Padeh Medical Center, Poria, Tiberias
  - Shamir Medical Center (Assaf Harofeh), Zrifin
- Italy (9):
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - A.O.U. di Ferrara, Ferrara, Emilia-Romagna
  - Asl Roma 6, Rome, Lazio
  - ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - IRCCS Istituto Clinico Humanitas - Humanitas Mirasole S.p.A., Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - IRCCS Fondazione Policlinico San Matteo, Pavia, Lombardy
  - A.O.U. di Sassari, Sassari, Sardinia
- Japan (21):
  - Seikeikai New Tokyo Heart Clinic, Matsudo, Chiba
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Matsuda Cardiovascular clinic, Sapporo, Hokkaido
  - National Hospital Organization Kobe Medical Center, Kobe, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Uji-Tokushukai Medical Center, Uji, Kyoto
  - Hirakata kohsai Hospital, Hirakata, Osaka
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - National Hospital Organization Hamada Medical Center, Hamada, Shimane
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni, Yamaguchi
  - Fukui Prefectural Hospital, Fukui
  - Okayama Rosai Hospital, Okayama
  - Osaka General Medical Center, Osaka
  - Toyama Prefectural Central Hospital, Toyama
- Malaysia (3):
  - Hospital Raja Perempuan Zainab II, Kelantan
  - Institute Jantung Negara, Kuala Lumpur
  - Sarawak Heart Centre, Sarawak
- Poland (9):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - 10 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ, Bydgoszcz
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - SPZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Uniwersyteckie Centrum Kliniczne Warszawskiego UM, Warsaw
  - IV Wojskowy Szpital Kliniczny z Poliklinika, SPZOZ, Wroclaw
  - Dolnoslaski Szp. Spec. im T.M. Centrum Medycyny Ratunkowej, Wroclaw
- Portugal (7):
  - Hospital de Cascais, Alcabideche, Lisbon District
  - CHTS - Hospital Padre Americo, Guilhufe, Porto District
  - CHS - Hospital Sao Bernardo, Setúbal, Setúbal District
  - Hospital Garcia de Orta, Almada
  - CHLO - Hospital Sao Francisco Xavier, Lisbon
  - Hospital da Luz - Lisboa, Lisbon
  - CHUP - Hospital Santo Antonio, Porto
- Russia (6):
  - Sci-Res. Institute of Complex Cardiovascular Disorders, Kemerovo
  - Research center of therapy and prophylactic medicine, Moscow
  - Moscow State University n.a. M.V. Lomonosov, Moscow
  - City hospital #15, Saint Petersburg
  - City Pokrovskaya Hospital, Saint Petersburg
  - Samara Regional Clinical Cardiology Dispensary n.a. Polyakov, Samara
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- South Africa (6):
  - Clinical Trial Systems, Pretoria, Gauteng
  - Durban Medical Centre, Durban, KwaZulu-Natal
  - Nash Ranjith Research Centre, Merebank, KwaZulu-Natal
  - TREAD Research cc, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Vergelegen Medi-Clinic, Somerset West, Western Cape
- Spain (9):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Ciutat Sanitària i Universitària de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Sant Joan Despi Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital Sanitas La Zarzuela, Aravaca, Madrid
  - Hospital Universitario Clinica Puerta de Hierro, Majadahonda, Madrid
  - Hospital Álvaro Cunqueiro, Babio - Beade, Pontevedra
  - Hospital del Mar, Barcelona
  - Hospital Virgen de la Victoria, Málaga
  - Complejo Hospitalario Ntra. Sra. de Valme, Seville
- Taiwan (4):
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei

REFERENCES:
- [Background] Butler J, Lam CSP, Anstrom KJ, Ezekowitz J, Hernandez AF, O'Connor CM, Pieske B, Ponikowski P, Shah SJ, Solomon SD, Voors AA, Wu Y, Carvalho F, Bamber L, Blaustein RO, Roessig L, Armstrong PW. Rationale and Design of the VITALITY-HFpEF Trial. Circ Heart Fail. 2019 May;12(5):e005998. doi: 10.1161/CIRCHEARTFAILURE.119.005998. PMID 31096775
- [Derived] deFilippi CR, Shah P, Shah SJ, Alemayehu W, Lam CSP, Butler J, Roessig L, O'Connor CM, Westerhout CM, Armstrong PW; VITALITY-HFpEF Study Group. Proteomics Identify Clinical Phenotypes and Predict Functional Outcomes in Heart Failure With Preserved Ejection Fraction: Insights From VITALITY-HFpEF. Circ Heart Fail. 2024 Sep;17(9):e011792. doi: 10.1161/CIRCHEARTFAILURE.124.011792. Epub 2024 Aug 29. PMID 39206547
- [Derived] Kaul P, Rathwell S, Lam CSP, Westerhout CM, Spertus JA, Anstrom KJ, Blaustein RO, Ezekowitz JA, Pieske B, Roessig L, Butler J, Armstrong PW; VITALITY-HFpEF Study Group. Patient-Reported Frailty and Functional Status in Heart Failure With Preserved Ejection Fraction: Insights From VITALITY-HFpEF. JACC Heart Fail. 2023 Apr;11(4):392-403. doi: 10.1016/j.jchf.2022.11.015. Epub 2023 Feb 1. PMID 36881394
- [Derived] Armstrong PW, Lam CSP, Anstrom KJ, Ezekowitz J, Hernandez AF, O'Connor CM, Pieske B, Ponikowski P, Shah SJ, Solomon SD, Voors AA, She L, Vlajnic V, Carvalho F, Bamber L, Blaustein RO, Roessig L, Butler J; VITALITY-HFpEF Study Group. Effect of Vericiguat vs Placebo on Quality of Life in Patients With Heart Failure and Preserved Ejection Fraction: The VITALITY-HFpEF Randomized Clinical Trial. JAMA. 2020 Oct 20;324(15):1512-1521. doi: 10.1001/jama.2020.15922. PMID 33079152
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 178 study centers worldwide, between 15-Jun-2018 (first subject first visit) and 04-Nov-2019 (last subject last visit).
Pre-assignment Details: Overall, 979 participants were screened, of whom 789 participants were randomized in the study. 788 of the randomized participants were allocated to study treatment, of whom 672 participants completed the study.
Groups:
- Vericiguat up to 10 mg: Participants received vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, with sham titration at week 6.
- Vericiguat up to 15 mg: Participants received vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, and to 15 mg at week 6 week.
- Placebo: Participants received placebo once daily and sham up-titration at weeks 2, 4, and 6.
Period: Overall Study
Arm/Group | Vericiguat up to 10 mg | Vericiguat up to 15 mg | Placebo
Started | 263 | 264 | 262
Treated | 262 | 264 | 262
Completed | 218 | 224 | 230
Not Completed | 45 | 40 | 32
Not completed — Adverse Event | 16 | 11 | 10
Not completed — Death | 11 | 7 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 3
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Withdrawal by Subject | 12 | 19 | 10
Not completed — Other | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: All participants randomized were valid for the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vericiguat up to 10 mg | Vericiguat up to 15 mg | Placebo | Total
Number analyzed (Participants) | 263 | 264 | 262 | 789
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (9.7) | 73.1 (9.1) | 72.8 (9.4) | 72.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 140 | 121 | 385
  Male | 139 | 124 | 141 | 404
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 21 | 23 | 72
  Not Hispanic or Latino | 235 | 242 | 238 | 715
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 4 | 11
  Asian | 24 | 26 | 25 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 9 | 21
  White | 228 | 224 | 222 | 674
  More than one race | 2 | 2 | 2 | 6
  Unknown or Not Reported | 1 | 1 | 0 | 2
Six-minute walk test [Mean (Standard Deviation); unit: Meters] — Six-minute walk test (6MWT) was conducted to test the physical limitations of the patient by assessing the patient's exercise capacity. The distance walked by the patient in 6 minutes was measured. FAS 6MWT: All patients randomized and treated (at least one dose of the study treatment), and who were able to perform at least one 6MWT assessment at both baseline and post-baseline (excluding safety follow-up). Population: The participants in FAS 6MWT were analyzed for this outcome measure.
  Meters
    number analyzed (Participants) | 236 | 245 | 240 | 721
    (all) | 292.13 (107.75) | 294.99 (118.00) | 295.80 (106.27) | 294.32 (110.72)
Kansas City Cardiopathy Questionnaire Physical limitation score (KCCQ PLS) [Mean (Standard Deviation); unit: Scores] — The KCCQ measures the impact of patients' heart failure, or its treatment, on 6 domains; Physical Limitation, Symptom (with subscores for frequency and burden), Quality of Life, Social Limitations, Symptom Stability and Self-Efficacy. Scores are calculated by summing domain responses and then transforming scores to a 0-100 unit scale with higher scores indicating better health status. FAS KCCQ: All patients randomized and treated (at least one dose of the study treatment), and had at least one observed KCCQ PLS assessment at both baseline and during post-baseline (excluding safety follow-up). Population: The participants in FAS KCCQ were analyzed for this outcome measure.
  Scores
    number analyzed (Participants) | 254 | 255 | 252 | 761
    (all) | 57.30 (24.77) | 60.03 (24.64) | 59.03 (24.00) | 58.79 (24.46)

OUTCOME MEASURES:

1. Primary Outcome: Change in KCCQ Physical Limitation Score From Baseline to Week 24
Description: The City Cardiomyopathy Questionnaire (KCCQ) measures the impact of patients' heart failure, or its treatment, on 6 domains; Physical Limitation, Symptom (with subscores for frequency and burden), Quality of Life, Social Limitations, Symptom Stability and Self-Efficacy. Scores are calculated by summing domain responses and then transforming scores to a 0-100 unit scale with higher scores indicating better health status.
Time Frame: From baseline to Week 24
Population: FAS KCCQ: All patients randomized and treated (at least one dose of the study treatment), and had at least one observed KCCQ PLS assessment at both baseline and during post-baseline (excluding safety follow-up) were valid for this analysis set.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Vericiguat up to 10 mg | Vericiguat up to 15 mg | Placebo
Number analyzed (Participants) | 254 | 255 | 252
Scores on a scale | 6.41 (1.592) | 5.47 (1.538) | 6.93 (1.535)
Statistical Analysis 1: Comparison: Vericiguat up to 10 mg vs Placebo; The analysis of each imputed dataset will be performed using mixed-effects model for repeated measures (MMRM), including treatment, region, heart rhythm, study visit as fixed effects, interaction between study visit and treatment group, and adjustment for the baseline PLS values as covariates; Test type: Other; p = 0.8008, Mixed model repeated-measures; Difference of LS-means = -0.52, 97.5% CI 2-sided [-5.17 to 4.13]
Statistical Analysis 2: Comparison: Vericiguat up to 15 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4722, Mixed model repeated-measures; Difference of LS-means = -1.46, 97.5% CI 2-sided [-6.02 to 3.10]

2. Secondary Outcome: Change in the Six-minute Walk Test (6MWT) From Baseline to Week 24
Description: 6MWT was conducted to test the physical limitations of the patient by assessing the patient's exercise capacity. The distance walked by the patient in 6 minutes was measured.
Time Frame: From baseline to Week 24
Population: FAS 6MWT: All patients randomized and treated (at least one dose of the study treatment), and who were able to perform at least one 6MWT assessment at both baseline and post-baseline (excluding safety follow-up) were valid for this analysis set.
Measure: Least Squares Mean (Standard Error); unit: Meters
Groups:
- Vericiguat up to 10 mg: Participants will receive vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, with sham titration at week 6.
- Vericiguat up to 15 mg: Participants will receive vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, and to 15 mg at week 6 week.
- Placebo: Participants will receive placebo once daily and sham up-titration at weeks 2, 4, and 6.
Arm/Group | Vericiguat up to 10 mg | Vericiguat up to 15 mg | Placebo
Number analyzed (Participants) | 236 | 245 | 240
Meters | 8.68 (5.841) | 5.00 (5.718) | 10.49 (5.512)
Statistical Analysis 1: Comparison: Vericiguat up to 10 mg vs Placebo; The analysis of each imputed dataset will be performed using mixed-effects model for repeated measures (MMRM), including treatment, region, heart rhythm, study visit as fixed effects, interaction between study visit and treatment group, and adjustment for the baseline 6MWT values as covariates; Test type: Other; p = 0.8054, Mixed model repeated-measures; Difference of LS-means = -1.81, 97.5% CI 2-sided [-18.30 to 14.67]
Statistical Analysis 2: Comparison: Vericiguat up to 15 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.4502, mixed model repeated measures; Difference of LS-means = -5.49, 97.5% CI 2-sided [-21.77 to 10.80]

3. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An AE is any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation patient after providing written informed consent for participation in the study. Adverse events are considered to be treatment-emergent if they have started or worsened after first application of study medication up to 5 calendar days after end of treatment with study medication.
Time Frame: From first application of study drug up to 5 calendar days after end of treatment with study drug
Measure: Number; unit: Participants
Arm/Group | Vericiguat up to 10 mg | Vericiguat up to 15 mg | Placebo
Number analyzed (Participants) | 262 | 264 | 262
Participants
  Any TEAE | 163 | 172 | 172
  Any study drug related TEAE | 38 | 42 | 24
  Any TESAE | 46 | 54 | 48

ADVERSE EVENTS:
Time Frame: Timeframe for reporting adverse events: From the first application of study medication up to 5 calendar days after end of treatment with study medication. Timeframe for number of death (all causes): After study medication start until last contact date. (The median follow-up time is 197 days.)
Groups:
- Vericiguat up to 10 mg: Subjects received vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, with sham titration at week 6.
- Vericiguat up to 15 mg: Subjects received vericiguat (BAY1021189) for 24 weeks, starting at 2.5 mg once daily at randomization and up-titrated to 5 mg at week 2, to 10 mg at week 4, and to 15 mg at week 6.
- Placebo: Subjects received placebo for 24 weeks, once daily, starting sham up-titration at weeks 2, 4, and 6.
Arm/Group | Vericiguat up to 10 mg | Vericiguat up to 15 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 15/262 | 10/264 | 7/262
Serious Adverse Events (participants affected / at risk) | 46/262 | 54/264 | 48/262
Other Adverse Events (participants affected / at risk) | 121/262 | 134/264 | 131/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat up to 10 mg (N=262) | Vericiguat up to 15 mg (N=264) | Placebo (N=262)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 4 (5) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 7 (7) | 4 (4)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Angiocardiogram (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3) | 4 (4)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 3 (3) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat up to 10 mg (N=262) | Vericiguat up to 15 mg (N=264) | Placebo (N=262)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 13 (13) | 9 (9)
Atrial fibrillation (Cardiac disorders) | 7 (8) | 7 (9) | 6 (6)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 4 (5) | 0 (0) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 1 (1) | 6 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 8 (9) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 6 (7) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (5) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 3 (4)
Chest pain (General disorders) | 2 (3) | 4 (4) | 3 (4)
Fatigue (General disorders) | 3 (4) | 7 (8) | 3 (3)
Oedema (General disorders) | 2 (2) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 16 (17) | 10 (13) | 8 (10)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 5 (5)
Bronchitis (Infections and infestations) | 3 (3) | 5 (6) | 7 (7)
Gastroenteritis (Infections and infestations) | 4 (5) | 5 (5) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 3 (4)
Nasopharyngitis (Infections and infestations) | 8 (9) | 7 (7) | 7 (7)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 6 (6) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7) | 4 (6)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (5) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 3 (4) | 0 (0)
Blood uric acid increased (Investigations) | 3 (3) | 4 (4) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 3 (3) | 2 (2)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 2 (2) | 1 (1) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (7) | 12 (13)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (7) | 8 (9) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 7 (8) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4) | 3 (4)
Dizziness (Nervous system disorders) | 8 (9) | 7 (9) | 11 (14)
Headache (Nervous system disorders) | 5 (6) | 6 (7) | 11 (16)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (2) | 3 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 4 (4) | 2 (2)
Renal impairment (Renal and urinary disorders) | 5 (6) | 4 (7) | 5 (7)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (4) | 7 (9)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (5) | 14 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 5 (5) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (5) | 6 (8)
Cataract operation (Surgical and medical procedures) | 1 (2) | 2 (2) | 3 (4)
Hypertension (Vascular disorders) | 5 (5) | 11 (12) | 10 (12)
Hypotension (Vascular disorders) | 16 (18) | 22 (31) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT03547583/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03547583/SAP_001.pdf